CLINICAL TRIAL: NCT05426889
Title: Establishment of a Clinical Efficacy Prediction System Based on the Role of Meningeal Lymphatic Vessels in the Absorption of Chronic Subdural Hematoma and Its Injury Mechanism
Brief Title: The Role of Meningeal Lymphatic Vessels in the Absorption of Chronic Subdural Hematoma and Its Injury Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022-0219
Record Dates: First submitted 2022-05-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Hematoma, Subdural, Chronic
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Other): undergo surgery
  Interventions: Procedure: subdural hematoma burr hole drainage
- non-surgical groups (Other): no surgery
  Interventions: Drug: drug conservative treatment

INTERVENTIONS:
Procedure: subdural hematoma burr hole drainage — For patients with larger hematoma, remove the hematoma by burr hole drainage
  Arms: Surgical
Drug: drug conservative treatment — The patient did not receive surgical treatment and chose conservative treatment
  Arms: non-surgical groups

SUMMARY:
Chronic subdural hematoma (CSDH) is a very common hemorrhagic disease of the nervous system, accounting for about 10% of hemorrhagic strokes. The incidence rate of elderly people over 65 years old is 58.1/100,000, and the incidence rate is increasing year by year, and it may reach 121/100,000 by 2030. At present, the specific pathogenesis of CSDH is still unclear. Although it has been clinically confirmed that a part of CSDH can be absorbed by itself, and some drugs such as atorvastatin can speed up the process, surgical treatments such as cranial craniotomy or cranial drilling hematoma removal are still the only options for patients with CSDH.

Lymphatic circulation spreads throughout most tissues of the human body, assists in removing metabolic wastes in the interstitium, maintains body fluid homeostasis, and plays a role in immune response and immune surveillance. For a long time, the central nervous system has been considered as an immune-privileged organ, that is, the central nervous system does not have the presence of the lymphatic system. Until 2015, Louveau et al. used immunofluorescence staining and other techniques to find functional lymphatic ducts adjacent to the dural venous sinuses in the mouse brain when looking for the channels for T cells to enter and leave the meninges, confirming the first intracranial meningeal lymphatic vessels. (mLVs), and found that mLVs express the classic markers of lymphatic endothelial cells (LECs), namely VEGFR3, prostate homeobox 1 (PROX 1), podoplanin, lymphatic endothelial markers transparent Ronidase receptor-1 (LYVE-1), etc. Relevant studies have confirmed that meningeal lymphatic vessels can drain interstitial fluid (ISF), macromolecular substances and immune cells out of the skull, providing a new drainage pathway for the excretion of metabolic waste from the central nervous system. Subsequent studies have confirmed that mLV is involved in the pathophysiological process of a series of neurological diseases such as Alzheimer's disease (AD), traumatic brain injury (TBI), and subarachnoid hemorrhage (SAH). This phenomenon suggests that mLVs play an important role in central nervous system diseases.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) is a very common hemorrhagic disease of the nervous system, accounting for about 10% of hemorrhagic strokes. The incidence rate of elderly people over 65 years old is 58.1/100,000, and the incidence rate is increasing year by year, and it may reach 121/100,000 by 2030. At present, the specific pathogenesis of CSDH is still unclear. Although it has been clinically confirmed that a part of CSDH can be absorbed by itself, and some drugs such as atorvastatin can speed up the process, surgical treatments such as cranial craniotomy or cranial drilling hematoma removal are still the only options for patients with CSDH. However, these surgical methods have a high recurrence rate of hematoma and the incidence of surgery-related complications, which brings a huge burden to the patient's family and society. Despite the presence of a large number of inflammatory cytokines in the CSDH content, only a minority of patients exhibited systemic inflammatory responses such as fever and increased white blood cell count during hematoma resorption. On the contrary, more CSDH patients showed a certain degree of neurological deficit symptoms, such as hemiplegia of one limb and cognitive function decline. These clinical phenomena have stimulated thinking about how CSDH is drained. If the hematoma is absorbed through the vascular system, why is no corresponding inflammatory response or clinical symptoms observed in CSDH patients. In addition, the cerebrospinal fluid (CSF) of patients with CSDH was clear and the cell count was within the normal range, indicating that CSDH did not flow into the CSF. Therefore, further exploring the drainage pathway of CSDH, understanding the absorption process and recurrence mechanism of CSDH, and developing new effective treatment methods are important issues faced by neurosurgery clinicians.

Lymphatic circulation spreads throughout most tissues of the human body, assists in removing metabolic wastes in the interstitium, maintains body fluid homeostasis, and plays a role in immune response and immune surveillance. For a long time, the central nervous system has been considered as an immune-privileged organ, that is, the central nervous system does not have the presence of the lymphatic system. Until 2015, Louveau et al. used immunofluorescence staining and other techniques to find functional lymphatic ducts adjacent to the dural venous sinuses in the mouse brain when looking for the channels for T cells to enter and leave the meninges, confirming the first intracranial meningeal lymphatic vessels. (mLVs), and found that mLVs express the classic markers of lymphatic endothelial cells (LECs), namely VEGFR3, prostate homeobox 1 (PROX 1), podoplanin, lymphatic endothelial markers transparent Ronidase receptor-1 (LYVE-1), etc. Relevant studies have confirmed that meningeal lymphatic vessels can drain interstitial fluid (ISF), macromolecular substances and immune cells out of the skull, providing a new drainage pathway for the excretion of metabolic waste from the central nervous system. Subsequent studies have confirmed that mLV is involved in the pathophysiological process of a series of neurological diseases such as Alzheimer's disease (AD), traumatic brain injury (TBI), and subarachnoid hemorrhage (SAH). This phenomenon suggests that mLVs play an important role in central nervous system diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis chronic subdural hematoma
* Hematoma thickness greater than 10mm on imaging

Exclusion Criteria:

* In patients with chronic subdural hematoma, only head CT examination was performed;
* There was previous brain injury (stroke, cerebral hemorrhage, etc., leaving relevant chronic changes on CT);
* Imaging data was lost and the onset of CSDH was accompanied by severe comorbidity disease patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance signal intensity of meningeal lymphatic vessels | The first day after admission
  The signal intensity of meningeal lymphatic vessels was measured by PACS system in hospital
Magnetic resonance signal intensity of meningeal lymphatic vessels | 3 days after surgery
  The signal intensity of meningeal lymphatic vessels was measured by PACS system in hospital
Magnetic resonance signal intensity of meningeal lymphatic vessels | 1 months after surgery
  The signal intensity of meningeal lymphatic vessels was measured by PACS system in hospital
Magnetic resonance signal intensity of meningeal lymphatic vessels | 6 months after surgery
  The signal intensity of meningeal lymphatic vessels was measured by PACS system in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated hosipital of zhejiang univerisity school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No